CLINICAL TRIAL: NCT04908878
Title: Analgesic Efficacy of Combined Ultrasound-Guided PECS II and Transeversus Thoracic Plane Blocks Versus Ultrasound-Guided Serratus Anterior Plane Block in Modified Radical Mastectomy: A Prospective Randomized Study
Brief Title: Combined PECS II and Transeversus Thoracic Plane Blocks Vs Serratus Anterior Plane Block in Modified Radical Mastectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Alshaimaa Soliman Alasrag, Resident at Anesthesiology, Surgical ICU and Pain medicine, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 33972/7/20
Record Dates: First submitted 2021-05-27; First posted 2021-06-01 (Actual); Last update posted 2022-11-29 (Actual); Status verified 2022-11

CONDITIONS: Ultrasound-Guided; Transeversus Thoracic Plane Blocks; Pectoral Nerve (PECS) Block; Serratus Anterior Plane Block; Modified Radical Mastectomy
MeSH Terms: conditions — Bites and Stings | interventions — thiamine triphosphorate; Dental Occlusion

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (pectoral nerve (PECS) block -transversus thoracic plane (TTP) block group) (Experimental): Patients will receive unilateral US-guided PECS II block and TTP block on the side of the operation after induction of general anesthesia.
  Interventions: Procedure: Pectoral nerve (PECS) block -transversus thoracic plane (TTP) block
- Group II (serratus anterior plane (SAP) block group) (Experimental): Patients will receive US-guided SAP block after induction of general anesthesia.
  Interventions: Procedure: Serratus anterior plane (SAP) block

INTERVENTIONS:
Procedure: Pectoral nerve (PECS) block -transversus thoracic plane (TTP) block — Patients will receive unilateral US-guided PECS II block and TTP block on the side of the operation after induction of general anesthesia.
  Arms: Group I (pectoral nerve (PECS) block -transversus thoracic plane (TTP) block group)
Procedure: Serratus anterior plane (SAP) block — Patients will receive US-guided SAP block after induction of general anesthesia.
  Arms: Group II (serratus anterior plane (SAP) block group)

SUMMARY:
The aim of this study is to evaluate the analgesic efficacy of combined ultrasound (US)-guided pectoral nerve (PECS) block II and transversus thoracic plane (TTP) block versus US-guided serratus anterior plane (SAP) block in female patients undergoing modified radical mastectomy.

ELIGIBILITY:
Inclusion Criteria:

* Female patients
* Aged 21-60 years
* ASA physical status I, II
* Scheduled for unilateral modified radical mastectomy

Exclusion Criteria:

1. Patient refusal.
2. Known hypersensitivity to local anesthetics.
3. Body mass index > 35 kg /m2.
4. Uncooperative or psychiatric patients.
5. Infection at the injection site.
6. Coagulation disorder.

Ages: 21 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — female
Enrollment: 70 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-06-02 (Actual)

PRIMARY OUTCOMES:
The total amount rescue analgesic consumption (morphine) in the first 24 hours postoperatively. | First 24 hours postoperatively.
  Rescue analgesia in the form of morphine (3mg IV) will be given if the VAS is ≥ 40, repeated with lock out interval of 5 min guided with the occurrence of complications till the VAS is decreased to less than 40.

SECONDARY OUTCOMES:
The degree of postoperative pain | First 24 hours postoperatively.
  Postoperative pain will be assessed by Visual Analog scale (VAS) on admission to Post-Anesthesia Care unit (PACU) and at 30 minutes and then 1,2,4,6,12,18 and 24 hours postoperative.
  VAS (0-100; where 0 represents no pain and 100 represents the worst pain).
Time to first rescue analgesia request. | First 24 hours postoperatively.
  Rescue analgesia in the form of morphine (3mg IV) will be given if the VAS is ≥ 40, repeated with lock out interval of 5 min guided with the occurrence of complications till the VAS is decreased to less than 40.
Intraoperative fentanyl consumption. | Intraoperative
  Additional boluses of fentanyl 0.5 µg /kg will be administered in case of inadequate analgesia that defined as increase of heart rate (HR) and /or mean arterial blood pressure (MAP) more than 20 % from baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine Tanta University, Tanta, Elgharbia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon reasonable request.
Supporting Information: Study Protocol, SAP
Time Frame: one year
Access Criteria: The data will be available upon reasonable request.